CLINICAL TRIAL: NCT03092050
Title: Group Therapy for Depressed Caregivers of Alzheimer's Disorder and Related Dementias
Brief Title: Group Therapy for Depressed Dementia Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Felipe A Jain, Psychiatrist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIT001; R21AG051970 (NIH)
Record Dates: First submitted 2017-03-10; First posted 2017-03-27 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Imagery, Psychotherapy; Mindfulness

STUDY DESIGN:
Intervention Model Description: 2 arm randomized controlled trial. During the conduct of the trial, the investigators noted that due to staffing constraints, participant availability, and funding limitations, it would not be feasible to complete a crossover study. This was due to the fact that the investigators were unable to offer crossover group therapy visits at the same time as the initial group sessions. Rather, groups with new participants had to be prioritized and scheduled during the most accessible time slots. Times that the investigators could offer for crossover groups were often inaccessible to participants. Thus, the investigators determined that in the context of this pilot trial, it was not feasible to conduct a full crossover trial due to accessibility. The trial design was therefore updated to parallel (in accordance with the initial funding application).
Who Masked: Participant
Masking Description: Participants were blinded to study hypotheses. Under UCSF IRB #16-20163, on 07.21.2016 (prior to participant enrollment), IRB approval was received for a single-blind study (participant blinding only) due to funding constraints.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facilitated Discussion (Active Comparator): Weekly facilitated discussion for 4 weeks
  Interventions: Behavioral: Facilitated Discussion
- Guided Imagery and mindfulness (Experimental): Weekly guided imagery and mindfulness for 4 weeks
  Interventions: Behavioral: Guided Imagery and Mindfulness

INTERVENTIONS:
Behavioral: Guided Imagery and Mindfulness — This is a behavioral intervention using guided imagery and mindfulness techniques.
  Arms: Guided Imagery and mindfulness
Behavioral: Facilitated Discussion — This is a behavioral intervention that involves discussion and group support.
  Arms: Facilitated Discussion

SUMMARY:
Depression in family caregivers of relatives with Alzheimer's Disorder and related dementias is a serious public health problem. This is a randomized, controlled, single-blind pilot clinical trial of depressed caregivers, to determine the efficacy and mechanisms of group therapy for depressed dementia caregivers.

DETAILED DESCRIPTION:
The trial was designed to measure clinical outcomes including depressive symptoms and other secondary outcomes of caregivers of persons living with dementia. It also included magnetic resonance imagery scanning at baseline (prior to study group) and post group to identify candidate mechanisms of effects.

Notes related to outcome measurement. On 05.10.2017 (prior to participant enrollment), all secondary outcomes were approved by the UCSF IRB #16-20163. It was noted in the IRB that the primary outcome timepoint was to be obtained 4 weeks after the first group session. Due to magnetic resonance imaging scanning scheduling constraints, which occurred at the same time as the 4 weeks visit, the outcome could not be exactly four weeks post the first group session but was collected approximately at this time.

On 05.10.2017 (prior to participant enrollment), three-month post group secondary outcomes were also approved.

ELIGIBILITY:
Inclusion Criteria:

Endorse clinically relevant baseline depressive symptoms Primary caregiver for a relative with dementia

Exclusion Criteria:

Age < 45 Meditation / guided imagery practice more than twice per week Ideas of harming relative with dementia Current violence towards relative with dementia Adult Protective Services report on file Primary psychiatric disorder other than unipolar major depression Cognitive impairment on the part of the caregiver (Mini Mental State Examination score less than 24) Unstable medical illness Planned surgery Active drug or alcohol abuse Inability to understand written and oral English.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Depression symptoms | approximately 4 weeks post initial group session
  Self reported depression symptoms (Quick Inventory of Depression Symptoms)

SECONDARY OUTCOMES:
Depression symptoms - moderate term | approximately 3 months post initial group session
  Self reported depression symptoms
Depression symptoms - clinician rated | approximately 4 weeks post initial group session and approximately 3 months post initial group session
  Hamilton Depression Rating Scale
Caregiver burden | approximately 4 weeks post initial group session and approximately 3 months post initial group session
  Caregiver Burden Scale self rated questionnaire
Anxiety symptoms | approximately 4 weeks post initial group session and approximately 3 months post initial group session
  State Trait Anxiety Inventory - Trait
Mindfulness | approximately 4 weeks post initial group session and approximately 3 months post initial group session
  Five Factor Mindfulness Questionnaire
Positive and Negative Affect | approximately 4 weeks post initial group session and approximately 3 months post initial group session
  Positive and Negative Affect Scale
Well-Being | approximately 4 weeks post initial group session and approximately 3 months post initial group session
  Mental Health Continuum Short Form
Stress | approximately 4 weeks post initial group session and approximately 3 months post initial group session
  Perceived Stress Scale
Resilience | approximately 4 weeks post initial group session and approximately 3 months post initial group session
  Connors Davidson Resilience Scale
Connectedness to Nature | approximately 4 weeks post initial group session and approximately 3 months post initial group session
  Connectedness to Nature Scale

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Jain, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States